CLINICAL TRIAL: NCT02427087
Title: Anthropometric Evaluation and Body Composition in Sedentary Postmenopausal Women With Nonalcoholic Fatty Liver Disease (NAFLD) Submitted to Physical Activity
Brief Title: Sedentary Postmenopausal Women With Nonalcoholic Fatty Liver Disease (NAFLD) Submitted to Physical Activity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Claudia Pinto Marques Oliveira, PhD, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 9022
Record Dates: First submitted 2015-03-04; First posted 2015-04-27 (Estimated); Last update posted 2015-04-27 (Estimated); Status verified 2015-04

CONDITIONS: Fatty Liver
Keywords: Nonalcoholic fatty liver; Physical activity; NAFLD; Anthropometry; Body Composition
MeSH Terms: conditions — Fatty Liver; Non-alcoholic Fatty Liver Disease; Motor Activity | interventions — Diet, Healthy

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Continuous Aerobic training (Active Comparator): Aerobic training continuous (n=19 patients) carry a protocol continuous aerobic training twice a week for 24 weeks and the session will last 60 minutes/2 days/week with recommendation for healthy diet.
  Interventions: Behavioral: Continuous Aerobic Training twice; Behavioral: Healthy Diet
- Healthy diet (Active Comparator): Diet group (n=21 patients) only recommendation for healthy diet.
  Interventions: Behavioral: Healthy Diet

INTERVENTIONS:
Behavioral: Continuous Aerobic Training twice — Supervised aerobic exercise program of 60 min/2 days/week at 60-85% of heart rate reserve for 24 weeks and healthy diet
  Arms: Continuous Aerobic training
Behavioral: Healthy Diet — Diet group (21) Recommendation for healthy diet.

SUMMARY:
Were included 40 patients with NAFLD followed at the Ambulatory of Non-alcoholic Fatty Liver Disease , Discipline of Clinical Gastroenterology, Clinic Hospital of the Medical School of the University of Sao Paulo (HC-FMUSP). Were included adults women of any race, aged 35 to 75 years, diagnosed with NAFLD and were followed for a period of six months. All patients underwent anthropometric and body composition, as well as analysis of clinical, laboratory before and after 6 months of exercise training protocol established.

The hypothesis of our research is that aerobic activity had a favorable impact on NAFLD. It is expected that the intervention of physical activity causes a decrease or no weight, decreased levels of aminotransferases, decreased insulin resistance assessed by homeostasis model assessment (HOMA) index and consequently decrease or reversal of hepatic steatosis.

DETAILED DESCRIPTION:
The Nonalcoholic fatty liver disease (NAFLD) is the most common form of liver diseases, affecting approximately 20-30% of the adult population and is more common in obese individuals (70-80%). The main risk factors associated with the disease are the components of the Metabolic syndrome. To date, there is no specific pharmacological treatment for NAFLD and changes in lifestyle with weight reduction and exercise are always recommended. Few data exist on the impact of physical activity and optimal nutritional strategy for the treatment of NAFLD. Seen the need to elucidate the impact of physical activity and the search for an ideal nutritional strategy in the treatment of NAFLD, the investigators proposed a randomized controlled trial evaluating the effects of a hypocaloric high-protein diet and aerobic exercise associated with this diet on metabolic and anthropometric parameters in sedentary postmenopausal women. 40 sedentary postmenopausal women with NAFLD who had liver biopsy for a period equal to or less than 2 (two) years were included. These patients were randomized into 2 groups: TRAINING group (19): aerobic training with hypocaloric high-protein diet and DIET group (21): only hypocaloric high-protein diet, and followed for a period of six months.

Laboratorial Assays (baseline and end of the protocol)

* AST, ALT, FA, GGT, albumine, Fe, fasting glucose, insulin, Total cholesterol, HDL, LDL, Triglycerides;
* TNFalfa, IL6, and adiponectin.

Anthropometrical Evaluation (baseline and end of the protocol)

* BMI, waist circumference, percent body fat, body fat mass, lean body mass

ELIGIBILITY:
Inclusion Criteria:

* 35-75 years of age, Female
* Biopsy-liver until 24 months previous that prove NAFLD or NASH
* Patients who agree to participate in the study and all signed informed consent.

Exclusion Criteria:

* Presence of alcoholism <20g (women) of ethanol/day, drugs, schistosomiasis, hepatitis B or C and other chronic liver diseases cause determined
* Without medical clearance for physical activity
* Without availability to attend appointments and physical activities 2x/week
* Significant change in dietary habits and/or exercise in the last 3 months that resulted in weight loss > 5%.

Ages: 35 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-01; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Efficacy in reduce inflammatory component of NASH for transient elastography liver | 6 months
  Determine the efficacy of the physical activity in reducing the systemic inflammatory component of NASH in patients with NAFLD for transient elastography liver, FibroScan (FS) [stiffness liver (SL) /CAP]

SECONDARY OUTCOMES:
Inflammatory systemic profile | 6 months
  Measure tumoral factor TNFalfa, interleukin 6 (IL6), adiponectin, lipidic and laboratory tests aspartate aminotransferase (AST), alanine aminotransferase (ALT), Cholesterol, total triglycerides, glicemy, insulin.

CONTACTS AND LOCATIONS:
Overall Officials: CLAUDIA PM MD OLIVEIRA, PhD, Principal Investigator — University of Sao Paulo, School of Medicine
Locations (1):
- University of Sao Paulo School of Medicine, São Paulo, São Paulo, Brazil